CLINICAL TRIAL: NCT02568241
Title: Interferon α After Prophylactic Donor Lymphocyte Infusion for the Relapse Prevention After Hematopoietic Stem Cell Transplantation
Brief Title: Interferon-α After DLI for the Prevention of Relapse
Acronym: IDPR-HSCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang, Principal Investigator, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-10
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Leukemia
Keywords: Interferon Alfa-2b; Relapse; Donor lymphocyte infusion
MeSH Terms: conditions — Leukemia; Recurrence | interventions — Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- interferon Alfa-2b (Experimental): High-risk acute leukemia patients after hematopoietic stem cell transplantation receive interferon Alfa-2b after prophylactic DLI
  Interventions: Other: Interferon Alfa-2b

INTERVENTIONS:
Other: Interferon Alfa-2b — High-risk acute leukemia patients receive prophylactic DLI at day 30-60 after hematopoietic stem cell transplantation,they received interferon α-2b (subcutaneously at dosages of 3 million units 2-3 times per week) . Interferon treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.
  Other Names: INF α-2b

SUMMARY:
This study aimed to evaluate the efficacy of interferon α after prophylactic donor lymphocyte infusion (DLI) among high-risk acute leukemia patients undergone unmanipulated blood and marrow transplantation. Hematopoietic stem cell transplantation (HSCT) is an effective treatment option for high-risk acute leukemia (AL). However, post-transplant relapse can occur in some patients, and the prognosis of these patients is usually very poor.Prophylactic DLI can decrease the risk of relapse of high-risk AL patients. Interferon α-2b exerts a relatively strong immunomodulatory effect. It can kill AL cells by regulating T-cell and/or natural killer cell functions.Consequently, interferon α-2b may have potential value for high-risk AL patients after transplantation. The study hypothesis: Using interferon α-2b after prophylactic DLI following hematopoietic stem cell transplantation in patients with high-risk AL can further reduce relapse rate and improve leukemia-free survival.

DETAILED DESCRIPTION:
High risk acute leukemia patients (except t(9;22)(q34; q11) cytogenetic abnormalities.) received interferon α-2b after prophylactic DLI at day 30-60 after unmanipulated blood and marrow transplantation. The end points were safety, leukemia-free survival, and immunologic response. Following time is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had high-risk acute leukemia after hematopoietic stem cell transplantation

Exclusion Criteria:

* Patients with t(9;22)(q34; q11) cytogenetic abnormalities;active graft-versus-host disease; active infection; organ failure, or relapse

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Leukemia free survival | Participants will be followed for an expected average of 3 years
  Number of participants survived without leukemia at three years

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun HUANG, MD, Principal Investigator — Peking University Institute of Hematology
Locations (1):
- Peking University Institute of Hematology,Beijing, Beijing, Beijing Municipality, China